CLINICAL TRIAL: NCT04257487
Title: Sulodexide (VESSEL®) for the Prevention of Recurrent Venous Thromboembolism in Elderly Patients After a First Episode of Venous Thrombembolism
Brief Title: Sulodexide, VESSEL®, for the Prevention of Recurrent Venous Thromboembolism (The Jason Study)
Acronym: Jason
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Arianna Anticoagulazione Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FAAI2.10.2018; 2019-000570-33 (EudraCT Number)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Venous Thromboembolism; Anticoagulant; Elderly
Keywords: Venous thromboembolism; Elderly; Sulodexide
MeSH Terms: conditions — Venous Thromboembolism | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subjects enrolled in the study, the experimenters, and the members of the Steering Committee, Adjudication Committee, Data Monitoring and Safety Board will not be aware of the assignment of the 3 treatments following their distribution.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment A (Active Comparator): Sulodexide (Vessel) 2 capsules of 250 LSU BID, for 12 months
  Interventions: Drug: Sulodexide
- Treatment B (Active Comparator): Sulodexide (Vessel) 1 capsule of 250 LSU and 1 indistinguishable placebo capsule BID., for 12 months
  Interventions: Drug: Sulodexide and placebo; Drug: Placebo
- Treatment C (Placebo Comparator): 2 indistinguishable placebo capsules BID, for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sulodexide — 2 soft capsules of Vessel® 250 LSU BID for 12 months
  Other Names: VESSEL®
  Arms: Treatment A
Drug: Sulodexide and placebo — 1 soft capsule of Vessel® 250 LSU and 1 soft capsule of placebo BID for 12 months
  Other Names: VESSEL® and placebo
  Arms: Treatment B
Drug: Placebo — Sugar pill manufactured to mimic sulodexide 250 LSU
  Other Names: 2 soft capsule of placebo BDI for 12 months
  Arms: Treatment B; Treatment C

SUMMARY:
The study aims at optimizing extended management of elderly patients (> 75 years) with at least one of the known bleeding risk factor, who suffered from first episode of venous thromboembolism of the lower extremity (proximal deep vein thrombosis with or without pulmonary embolism) (VTE). Patients were randomized to receive three different treatment: Sulodexide 250 mg BIS in die; Sulodexide 500 BID in die or indistinguishable placebo to verify the efficacy and safety of extended treatment for 12 months with Sulodexide (Vessel®) in the secondary prevention of Deep Vein Thrombosis / Pulmonary Embolism (DVT/PE) recurrence.

DETAILED DESCRIPTION:
This prospective cohort study aims to assess the efficacy and safety of the extended treatment with Sulodexide (Vessel®) in the secondary prevention of DVT / PE recurrence in elderly outpatients (≥ 75 years old at the time of inclusion) ), with at least one of the known bleeding risk factor, who had a first episode of lower extremity proximal DVT and / or PE, idiopathic or associated with weak or removed risk factors, and who have received standard treatment with any oral anticoagulant drug lasting at least 3 months. The study seeks to verify the safety of the Sulodexide therapy, demonstrating non-inferiority compared to placebo, with an incidence of major bleeding around 1% (upper confidence limit not > 3%).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a first event of proximal lower extremity DVT and / or PE, idiopathic or associated with weak or removed risk factors.
2. Patients aged ≥75 years at the time of enrolment
3. Patients with at least one of the known risk factors of bleeding (APPENDIX 1):

   1. Hypertension
   2. Renal failure
   3. Thrombocytopenia
   4. Diabetes
   5. Antiplatelet therapy (ASA maximum 140 mg/die)
   6. Frequent falls (>2 /years)
   7. Nonsteroidal anti-inflammatory drug
   8. Liver failure
   9. Previous Stroke
   10. Anemia
   11. Poor anticoagulant control
   12. Alcohol abuse
4. Patients of both sexes.
5. Patients who at the time of enrolment have already undergone a period of anticoagulant therapy (AT, with any medication) of at least 3 months and the therapy has not been suspended for more than 30 days.
6. Patients with no other AT indications.
7. Patients capable and able to provide informed consent

Exclusion Criteria:

1. Patients aged <75 years at the time of the recruitment visit.
2. "Provoked" index event, which occurred:

   * Within 3 months of surgery or major trauma,
   * Bed Rest > 4 days,
   * Cast / immobility within 3 months.
3. Index event represented by severe PE, with life threatening risk or treated with thrombolytic therapy.
4. Index event represented by isolated distal DVT or superficial venous thrombosis.
5. Thrombotic event in sites other than the deep proximal veins of the lower limbs.
6. Anticoagulant therapy for less than 3 months at the time of enrolment.
7. Discontinuation of anticoagulant therapy for over thirty days at the time of enrolment
8. Recurrent episodes of DVT ± PE

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1455 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Number and rate of patients with confirmed recurrent VTE and VTE-related death (efficacy). | From date of enrollment until the date of first documented event assessed up to 12 months
  The occurrence of proximal deep vein thrombosis with or without pulmonary embolism (new or recurrent episode) wil be recorded in all patients
Number and rate of major Bleeding events (defined according to International Society on Thrombosis and Haemostasis guidelines (safety) | From date of enrollment until the date of first documented event assessed up to 12 months
  Fatal bleeding; intracranial; intraspinal; intraocular; pericardial; intra-articular; intramuscular with compartment syndrome; retroperitoneal,; acute clinically overt bleeding will be recorded in all patients

SECONDARY OUTCOMES:
Number of and rate of thromboembolic events | From date of enrollment until the date of first documented event assessed up to 12 months
  Transient ischemic attack (TIA), Stroke, Myocardial infarction will be recorded in all patients
Presence of severe post-thrombotic syndrome according to Villalta Score | 12 months
  Patient with deep vein thrombosis as index event will be evaluated, at the and of follow-up, applying Villalta score, commonly used to diagnose post-thrombotic syndrome in the subacute phase of thrombosis. The presence of venous ulcer of the leg or a score > of 15 points indicate the occurrence of severe post-thrombotic syndrome. The maximum score is 33. The score from 5 to 9 points indicate mild post-thrombotic syndrome and from 10 to 15 points indicate moderate post-thrombotic syndrome
Number and rate of non major bleeding complications | From date of enrollment until the date of first documented event assessed up to 12 months
  In all patients will be recorded any sign or symptom of hemorrhage that does not fit the criteria for the definition of major bleeding but does meet at least one of the following criteria: 1)requiring medical intervention by a healthcare professional; 2) leading to hospitalization or increased level of care;3) prompting a face to face evaluation
Number and rate of dead patients (overall mortality) | From date of enrollment until the date of first documented event assessed up to 12 months
  VTE-related death; cardiovascular related-death; bleeding-related death; death for: cancer, infectious disease and unknown cause; sudden death will be recorded in all patients

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Lodigiani, MD,PhD, Study Chair — IRCCS Humanitas, Rozzano (Milano)
Locations (1):
- Corrado Lodigiani, Rozzano, Italy

REFERENCES:
- [Derived] Palareti G, Legnani C, Antonucci E, Zorzi S, Bignamini AA, Lodigiani C, Tosetto A, Bertu L, Pengo V, Testa S, Ageno W, Prisco D, Prandoni P, Poli D. Design and rationale of a randomized, placebo-controlled trial on the efficacy and safety of sulodexide for extended treatment in elderly patients after a first venous thromboembolism. Intern Emerg Med. 2021 Mar;16(2):359-368. doi: 10.1007/s11739-020-02381-5. Epub 2020 May 25. PMID 32451933

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04257487/Prot_SAP_000.pdf